CLINICAL TRIAL: NCT00005847
Title: A Randomized Phase II Trial of Mitoxantrone, Estramustine and Navelbine or 13-cis Retinoic Acid, Interferon and Paclitaxel in Patients With Metatstatic Hormone Refractory Prostate Cancer
Brief Title: Chemotherapy With or Without Biological Therapy in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067865; E-3899
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interferon-alpha; Estramustine; Isotretinoin; Mitoxantrone; Paclitaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: estramustine phosphate sodium
Drug: isotretinoin
Drug: mitoxantrone hydrochloride
Drug: paclitaxel
Drug: vinorelbine ditartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. It is not yet known which treatment regimen is more effective in treating metastatic prostate cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of combination chemotherapy with that of chemotherapy plus biological therapy in treating patients who have progressive or metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of estramustine, mitoxantrone, and vinorelbine vs isotretinoin, interferon alfa, and paclitaxel on PSA response in patients with metastatic hormone-refractory prostate cancer.
* Determine the toxic effects of each regimen in this patient population.
* Determine the effect of each regimen on pain, fatigue, and quality of life in these patients.
* Determine the objective response rate among the subset of patients who have bidimensionally measurable disease to each regimen after treatment.
* Determine the effect of each regimen on peripheral blood mononuclear cell BCL-2 in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease (measurable vs nonmeasurable and elevated PSA). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive vinorelbine IV over 10 minutes on days 2 and 9 followed by mitoxantrone IV over 10 minutes on day 2 only. Oral estramustine is administered every 12 hours on days 1-5. Courses repeat every 3 weeks in the absence of unacceptable toxicity, disease progression, or administration of the maximum cumulative dose of mitoxantrone.
* Arm II: Patients receive oral isotretinoin and interferon alfa subcutaneously on days 1 and 2 and paclitaxel IV over 1 hour on day 2 weekly for 6 weeks. Courses repeat every 8 weeks in the absence of unacceptable toxicity or disease progression.

Quality of life is assessed at baseline, on day 2 of courses 2, 4, and 6 (arm I), on day 22 of course 1 and day 1 of courses 2 and 3 (arm II), and then at completion of treatment.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 70-114 patients (35-57 per arm) will be accrued for this study within 14-23 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Evidence of progressive metastatic disease (e.g., bone, pelvic mass, lymph node, liver or lung metastases)

  * Radiologic evidence of hydronephrosis only does not constitute evidence of metastatic disease
* Must not have an elevated serum alkaline phosphatase or PSA level as only evidence of disease
* If bone metastases only (i.e., lacking soft tissue disease), must have PSA level of at least 20 ng/mL
* If soft tissue metastases and/or visceral disease, must have either bidimensionally measurable disease or PSA level of at least 20 ng/mL
* Must have had prior bilateral orchiectomy or other primary hormonal therapy (e.g., estrogen therapy or LHRH blocker plus flutamide) with evidence of treatment failure
* No carcinomatous meningitis or brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* See Disease Characteristics
* Bilirubin no greater than 1.5 mg/dL
* SGOT/SGPT no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No active angina pectoris
* No New York Heart Association class III or IV heart disease
* No myocardial infarction within the past 6 months
* No deep venous thrombosis
* LVEF at least 50% by MUGA

Other:

* Fertile patients must use effective contraception during and for 1 month after study
* Prior malignancy allowed provided curatively treated and disease free for appropriate time period for specific cancer
* No other serious medical illness or active infection that would preclude protocol therapy
* No concurrent prolonged exposure to sunlight
* No concurrent alcohol consumption

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy, including neoadjuvant chemotherapy or single-agent estramustine

Endocrine therapy:

* See Disease Characteristics
* If no prior bilateral orchiectomy, must continue LHRH agonist therapy (e.g., depot leuprolide or goserelin)
* At least 4 weeks since prior flutamide or flutamide with evidence of progressive disease
* At least 6 weeks since prior bicalutamide with evidence of progressive disease

Radiotherapy:

* More than 4 weeks since prior radiotherapy
* No prior strontium chloride Sr 89, samarium Sm 153 lexidronam pentasodium, or other radioisotope therapies

Surgery:

* See Disease Characteristics

Other:

* Recovered from all toxic effects due to prior treatment for prostate cancer
* No concurrent milk, milk products, antacids, calcium-containing drugs, or any food with estramustine (arm I only)
* No concurrent vitamin supplements containing vitamin A (arm II only)

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04-05 (Actual); Primary Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. DiPaola, MD, Study Chair — Rutgers Cancer Institute of New Jersey; Robert G. Kilbourn, MD, PhD, Study Chair — Texas Oncology, PA - San Marcos
Locations (19):
- United States (19):
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Tufts - New England Medical Center, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Dipaola RS, Manola J, Li S, et al.: A randomized phase II trial of mitoxantrone, estramustine and vinorelbine or 13-cis retinoic acid, interferon and paclitaxel in patients with metastatic hormone refractory prostate cancer: results of ECOG 3899. [Abstract] J Clin Oncol 22 (Suppl 14): A-4594, 405s, 2004.